CLINICAL TRIAL: NCT03793140
Title: A Phase II Clinical Trial of CPI-613 in Patients With Relapsed or Refractory Burkitt Lymphoma/Leukemia or High-grade B-cell Lymphoma With Rearrangements of MYC and BCL2 and/or BCL6
Brief Title: A Study of CPI-613 for Patients With Relapsed or Refractory Burkitt Lymphoma/Leukemia or High-Grade B-Cell Lymphoma With High-Risk Translocations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: City of Hope Medical Center (Other); Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other); George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-443
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Leukemia
Keywords: Burkitt Lymphoma/Leukemia; high-grade B-cell lymphoma; CPI-613
MeSH Terms: conditions — Lymphoma; Leukemia; Burkitt Lymphoma | interventions — devimistat

STUDY DESIGN:
Intervention Model Description: This is an open-label multicenter, single-arm, phase II trial of CPI-613 monotherapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 (Experimental): CPI-613 IV induction (Days 1-5 for first 2 Cycles [14-day cycles]), followed by CPI-613 IV maintenance (Days 1-5 for all Cycles thereafter [21-day cycles].
  Interventions: Drug: CPI-613

INTERVENTIONS:
Drug: CPI-613 — CPI-613 [2,500 mg/m2/day IV] over 2 hours (+/- 10 mins) Induction tx: Cycle 1 and 2: Treatment on Days 1-5 (Each cycle is 14 days). (Each Cycle is 14 days) Maintenance tx: All subsequent Cycles: Treatment with CPI-613 [2,500 mg/m2/day IV] over 2 hours (+/- 10 mins) on Days 1-5 (Each Cycle is 21 days)

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug, CPI-613.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 12 years of age.
* Histologic diagnosis of Burkitt Lymphoma/Leukemia or high-grade B-cell lymphoma with rearrangements of MYC and BCL2 and/or BCL6 confirmed at enrolling institution or plasmablastic lymphoma or high-grade B-cell lymphoma with rearrangements of MYC without bcl-2
* Failure of at least one previous line of therapy.
* Failure after prior bone marrow transplant, or ineligible for or opted not to participate in bone marrow transplantation for Burkitt Lymphoma/Leukemia, or DHL/THL.
* ECOG Performance Status of ≤ 3.

  1. For patients less than 16 years of age, Lansky score ≥ 30
  2. For patients 16- 17 years of age, Karnofsky score ≥ 30
* Measurable disease as defined RECIL criteria (2017) or isolated bone marrow involvement.
* Patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with anti-cancer drugs, radiotherapy or other anti-cancer modalities. Patients with persistent, non-hematologic, non-infectious toxicities from prior treatment must have documented resolution to ≤ Grade 2.
* Patients must have, or be willing and eligible to undergo placement of, a working central venous access device
* Venous access available (e.g., portacath, PICC line or equivalent).
* Laboratory values obtained ≤ 2 weeks prior to enrollment must demonstrate adequate hepatic function, renal function, and coagulation as defined below:

  * Aspartate aminotransferase (AST/SGOT) ≤ 5x upper normal limit (ULN)
  * Alanine aminotransferase (ALT/SGPT) ≤ 5x ULN
  * Total bilirubin ≤1.5x ULN (unless related to hemolysis or Gilbert's syndrome, or involvement by lymphoma; if involvement by lymphoma: total bilirubin </= 3.0 x ULN)
  * Creatinine clearance >=40cc min either by 24-hour creatinine clearance or calculated from the modified Cockcroft-Gault equation (with the use of ideal body mass [IBM] instead of mass): CRCL =(140-Age) × IBM (kg) × [0.85 if female]/[(72 • serum creatinine (mg/dL)]
  * For patients less than 16 years of age, the Bedside Schwartz equation or Creatinine-Cystatin C-based CKiD equation should be used for creatinine-based GFR calculation
  * International Normalized Ratio (INR) must be <1.5. Due to the occurrence of thrombocytopenia, patients should not enter with coagulopathy. Patients on anticoagulants should be on short-acting therapy (e.g. low molecular weight heparin) rather than oral anticoagulants.
  * Albumin ≥2.0 g/dL (or ≥20 g/L)
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study and must have a negative serum or urine pregnancy test within 2 weeks prior to treatment initiation.
* Females must agree to abstain from breastfeeding during study participation
* Fertile men must practice effective contraceptive methods during the study unless documentation of infertility exists.

Exclusion Criteria:

* Patients that have received a chemotherapy regimen with stem cell support in the previous 2 months.
* Any medical condition that is clinically unstable despite present therapy (i.e. uncontrolled infection).
* Platelets < 50,000/mm3 unless attributable to marrow based (either Burkitt lymphoma or DHL/THL.) Note: Patients with leukemia/lymphoma in the marrow 25,000-50,000 will be assessed for grade 4 thrombocytopenia unless they have platelet recovery above grade 3. Patients entering with platelets <25,000 will only be assessed for thrombocytopenia related to drug if they recover to grade 3 or higher.
* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, coronary artery disease, myocardial infarction within the past 3 months, uncontrolled cardiac arrhythmia, pericardial disease or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patient's risk for toxicity.
* Patients with active central nervous system (CNS) parenchymal disease. Patients with leptomeningeal disease are allowed as long as the CSF has cleared for more than 4 weeks and the patient is receiving maintenance intrathecal/intra Ommaya therapy.
* Any active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any condition or abnormality which may, in the opinion of the investigator, compromise his or her safety.
* HIV patients with any of the following: a) uncontrolled HIV infection defined as an HIV viral load > 100K copies/mL, b) a documented opportunistic infection within the last 90 days, c) concurrent HIV therapy with zidovudine or any strong CYP3A4 inhibitor (e.g. ritonavir or cobicistat) within 7 days of study drug due to potential drug-drug interaction.
* Patients who have received radiotherapy, surgery, treatment with cytotoxic agents, treatment with biologic agents, immunotherapy , or any other anti-cancer therapy for any kind for cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of CPI-613 treatment with the exclusion of radiation to one area (e.g. whole brain or involved nodal site) that does not interfere with response assessment in other sites. A course of steroids (up to 14 days total) prior to study initiation is acceptable.
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.
* Prior allogeneic stem cell transplant within 2 months of study start

  1. Patients with active graft-versus-host-disease are not eligible
  2. Patients receiving immunosuppressive therapy for prevention of graft-versus-host disease are not eligible

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate of CPI-613 | 3 years
  ORR will be defined as rate of complete response (CR) + partial response (PR) + minor response (MR) + Stable disease (SD) as determined as per the RECIL criteria. RECIL criteria for response assessment in lymphoma and/or bone marrow biopsy (depending on sites of disease as indicated by treating physician).

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Noy, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Steiner R, Nikolaenko L, Nair R, Seshan V, Thiruvengadam SK, Khan N, Abramson JS, Horwitz S, Matasar M, Owens C, Rodriguez Rivera II, Straus DJ, Pardee TS, Luther S, Saboukoulou S, Thet WS, Vemuri S, Noy A. Novel devimistat results in complete remissions in heavily pretreated Burkitt lymphoma in a phase 2 trial. Blood Adv. 2025 Nov 11;9(21):5556-5563. doi: 10.1182/bloodadvances.2025016168. PMID 40674734
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm